CLINICAL TRIAL: NCT03777228
Title: Integrated Eye Tracking and Neural Monitoring for Enhanced Assessment of Mild TBI: Primary Study
Status: Completed | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: G172NU-S1
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2017-06

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Traumatic brain injury, concussion, eye tracking, EEG, fMRI, DTI, Neurocognition
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Control: Individuals without traumatic brain injury
- Mild TBI: Individuals with mild traumatic brain injury
- Moderate to Severe TBI: Individual with moderate to severe traumatic brain injury

SUMMARY:
This study was conducted to develop and validate integrated eye tracking and EEG measures for assessment of mild traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* age 18 -55, ability to use left and right hands and right foot to complete cognitive and motor tasks without adaptive equipment, and fluent in English

Exclusion Criteria:

* history of severe TBI, history of neurological illness unrelated to TBI, vision problems that are uncorrected by contacts or glasses, history of psychotic disorder, or current homicidal or suicidal ideation or intent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited through USUHS, the Walter Reed National Military Medical Center, the National Intrepid Center of Excellence, Malcolm Grow Medical Center, the Washington DC VA Medical Center, VA outpatient treatment centers and Vet Centers in the greater Washington, D.C. area, Fort Belvoir, Fort Detrick and Fort Meade, public areas in the surrounding community, and in clinical settings such as such as concussion clinics, neurorehabilitation centers, and other local private practices.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Saccadic RT | 1 day (single time point)
  Saccadic Response Time